CLINICAL TRIAL: NCT05520112
Title: Treatment of Recurrent Pregnancy Loss Using Mesenchymal Stem Cells Capable of Differentiation in the Endometrial-decidual Direction
Brief Title: Treatment of Recurrent Pregnancy Loss Using Mesenchymal Stem Cells
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Institute of Biophysics and Cell Engineering of National Academy of Sciences of Belarus (Other Government)
Collaborators: Belarusian Medical Academy of Post-Graduate Education (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IBCE_MSC(Endometrial)
Record Dates: First submitted 2022-08-26; First posted 2022-08-29 (Actual); Last update posted 2022-08-29 (Actual); Status verified 2022-08

CONDITIONS: Recurrent Pregnancy Loss
Keywords: Recurrent Pregnancy Loss, Mesenchymal stem cells

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patients with Recurrent Pregnancy Loss receiving standard treatment and autologous MSC (Experimental): Experimental: Patients with Recurrent Pregnancy Loss receiving standard treatment and autologous MSC
  Interventions: Biological: Mesenchymal stem cells capable of differentiation in the endometrial-decidual direction; Other: Standard treatment according to the clinical protocols
- Standard treatment according to the clinical protocols (Active Comparator): Standard treatment of Recurrent Pregnancy Loss according to the clinical protocols
  Interventions: Other: Standard treatment according to the clinical protocols

INTERVENTIONS:
Biological: Mesenchymal stem cells capable of differentiation in the endometrial-decidual direction — Mesenchymal stem cells capable of differentiation in the endometrial-decidual direction
  Arms: Patients with Recurrent Pregnancy Loss receiving standard treatment and autologous MSC
Other: Standard treatment according to the clinical protocols — Standard treatment of Recurrent Pregnancy Loss according to the clinical protocols

SUMMARY:
Treatment of Recurrent pregnancy loss using mesenchymal stem cells capable of differentiation in the endometrial-decidual direction.

DETAILED DESCRIPTION:
Treatment of Recurrent pregnancy (characterized by the presense of thin endometrium) loss using mesenchymal stem cells capable of differentiation in the endometrial-decidual direction.

ELIGIBILITY:
Inclusion Criteria:

* female patients of reproductive age 18-49 years;
* recurrent pregnancy loss without current pregnancy with thin endometrium;
* unsuccessful IVF cycles due to thin endometrium;
* endometrial thickness is ≤6 mm in the first and second phases of the menstrual cycle;
* uterine infertility associated with endometrial hypoplasia;
* the absence of genetic diseases that prevent pregnancy;
* absence of taking hormonal drugs for 3 months prior to enrollment in the study.

Exclusion Criteria:

* patients with congenital malformations of the genital organs: agenesis and aplasia of the uterus, bicornuate uterus, unicornuate uterus, congenital fistula between the uterus and the digestive and urinary tracts, other congenital anomalies of the body and cervix. congenital anomaly of the body and cervix, unspecified, other specified developmental anomalies;
* acute inflammatory processes in the uterus;
* acute or chronic infectious and non-infectious diseases in the acute stage, including HIV, hepatitis B and C, syphilis, tuberculosis, chlamydia, myco-, ureaplasmosis, herpes, toxoplasmosis, rubella, cytomegalovirus, gonorrhea, trichomoniasis, etc.;
* autoimmune diseases;
* patients with malignant tumor including a history;
* patients with benign tumors of the uterus and appendages;
* miscarriage not associated with a thin endometrium, including immunological origin;
* hyper- or hypogonadotropic insufficiency of ovarian function, hyperandrogenemia of any origin;
* allergic reactions in the acute stage, established hypersensitivity to any component of the biomedical cell product;
* permanent therapy with cytostatics, hormones;
* mental and behavioral disorders that make it impossible for patients to participate in the study, drug and/or alcohol addiction.

Ages: 18 Years to 49 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2022-11-01 (Estimated); Primary Completion 2023-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Adverse effects associated with the therapy | 1 year
  Determination of adverse effects associated with the therapy
Adverse effects associated with the therapy | 1 month
  Determination of adverse effects associated with the therapy
Percent of patients with successful pregnancy | 1 year
  Percent of patients with successful pregnancy within 1 year after treatment

CONTACTS AND LOCATIONS:
Overall Officials: Andrei Hancharou, Dr, Study Chair — Institute for biophysics and cellular engineering NAS of Belarus
Locations (1):
- Institute of Biophysics and Cell Engineering of National Academy of Sciences of Belarus, Minsk, Belarus

IPD SHARING:
Plan to Share IPD: No